CLINICAL TRIAL: NCT03804060
Title: A Multicenter, Prospective, Randomized-controlled Trial to Assess the Safety and Feasibility of Cooling as an Adjunctive Therapy to Thrombectomy and Reperfusion in Patients With Acute Cerebral Ischemia and Stroke
Brief Title: REperfusion With Cooling in CerebraL Acute IscheMia II
Acronym: RECCLAIM-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZOLL Circulation, Inc., USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDC-3599
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Stroke
Keywords: Therapeutic Hypothermia; Cooling; Stroke; Neurological Acute Care
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cooling + Recanalization (Experimental): The subjects will be considered to be enrolled in the Test Arm of the trial when all inclusion and exclusion criteria have been met, the informed consent form has been signed, and randomization to the Test Arm of the trial to allow cooling with the Thermogard XP3 IVTM System before and after recanalization.
  Interventions: Device: Thermogard XP3
- Recanalization only (Active Comparator): The subjects will be considered to be enrolled in the Control Arm of the trial when all inclusion and exclusion criteria have been met, the informed consent form has been signed, and randomization to the Control Arm of the trial to allow recanalization only.
  Interventions: Procedure: Recanalization only

INTERVENTIONS:
Device: Thermogard XP3 — Cooling with the ZOLL® Circulation catheter and the ZOLL® Intravascular Temperature Management system to initiate and maintain hypothermia for 6 hours as an adjunct to endovascular Recanalization.
  Arms: Cooling + Recanalization
Procedure: Recanalization only — Standard of Care for recanalization
  Arms: Recanalization only

SUMMARY:
The primary objective of this study is to determine the feasibility and safety of achieving rapid hypothermia with the Proteus Intravascular Temperature Management (IVTM) system for patients experiencing acute ischemic stroke due to a large vessel occlusion.

ELIGIBILITY:
All Inclusion Criteria must be answered YES for Patient to be eligible.

1. Age ≥18 and ≤85;
2. Signs and symptoms consistent with an acute ischemic stroke with anterior circulation large vessel occlusion (M1 MCA, carotid-terminus occlusion, Tandem occlusion allowed (Extracranial ICA+carotid T or M1 MCA)) as determined by CT imaging; (i.e., hyperdense sign on non-contrast CT or CT angiogram);
3. Ability to perform arterial puncture within 24 hours from symptom onset or LKN;
4. ASPECTS score of 6-10 on non-contrast CT of the brain if under 80 years; ASPECTS 9-10 if age 80-85;
5. For transfer patients with anticipated arterial puncture greater than 6 hours from symptom onset or LKN, qualifying imaging must be performed within 2 hours prior to enrolling hospital arrival; or with a newly obtained non-contrast CT scan if this time is exceeded
6. Candidate for endovascular thrombectomy therapy in accordance with best practices per AHA standard stroke guidelines meeting all labeling requirements for EVT in the trial;
7. No contraindications to general anesthesia, conscious sedation or allergies to any components associated with the anticipated diagnostic or treatment procedures that cannot be treated;
8. A pre-stroke modified Rankin Score (mRS) of 0 or 1 (Appendix 4);
9. Baseline CT scan shows no hemorrhage;
10. NIHSS greater than or equal to 8 (Appendix 3);
11. Patient is capable of complying with study procedures and agrees to complete all required study procedures, study visits and associated activities;
12. Legally authorized representative must be able to understand and give written informed consent. Patient will assent if capable. Patient may be re-consented once it is established that there is no memory loss or cognitive impairment.

5.2 Exclusion Criteria In order to be eligible for participation, patients must meet all Inclusion and Exclusion Criteria.

Inclusion Criteria All Inclusion Criteria must be answered YES for Patient to be eligible.

1. Age ≥18 and ≤85;
2. Signs and symptoms consistent with an acute ischemic stroke with anterior circulation large vessel occlusion (M1 MCA, carotid-terminus occlusion, Tandem occlusion allowed (Extracranial ICA+carotid T or M1 MCA)) as determined by CT imaging; (i.e., hyper dense sign on non-contrast CT or CT angiogram);
3. Ability to perform arterial puncture within 24 hours from symptom onset or LKN;
4. ASPECT score of 6-10 on non-contrast CT of the brain if under 80 years; ASPECTS 9-10 if age 80-85;
5. For transfer patients with anticipated arterial puncture greater than 6 hours from symptom onset or LKN, qualifying imaging must be performed within 2 hours prior to enrolling hospital arrival or with a newly obtained non-contrast CT scan if this time is exceeded;
6. Candidate for endovascular thrombectomy therapy in accordance with best practices per AHA standard stroke guidelines meeting all labeling requirements for EVT in the trial;
7. No contraindications to general anesthesia, conscious sedation or allergies to any components associated with the anticipated diagnostic or treatment procedures that cannot be treated;
8. A pre-stroke mRS of 0 or 1 (Appendix 4);
9. Baseline CT scan shows no hemorrhage;
10. NIHSS greater than or equal to 8 (Appendix 3);
11. Patient is capable of complying with study procedures and agrees to complete all required study procedures, study visits and associated activities;
12. Legally authorized representative must be able to understand and give written informed consent. Patient will assent if capable. Patient may be re-consented once it is established that there is no memory loss or cognitive impairment.

Exclusion Criteria All Exclusion Criteria must be answered NO to be eligible.

1. Patient arrives to the enrolling hospital intubated
2. Female patients of childbearing potential who are known to be or may be pregnant;
3. The patient has a known history of bleeding diathesis, coagulopathy, cryoglobulinemia, sickle cell anemia, will refuse blood transfusions or contraindication to heparin; history of genetically confirmed hypercoagulable syndrome
4. The patient has a height of < 1.5 meters (4 feet 11 inches);
5. Use of warfarin with INR > 1.7;
6. Blood clinical chemistry potassium (K+) < 2.7;
7. History of severe dementia and currently taking medication for cognitive impairment or behavior disorder;
8. End stage renal disease on hemodialysis;
9. Known presence of an IVC filter;
10. Contrast dye allergy with history of anaphylaxis, known serious sensitivity to contrast agents or any condition in which angiography is contraindicated;
11. Known to have contraindications to radiological imaging;
12. Known allergy to meperidine or buspar or dexmedetomidine;
13. Sustained hypertension (SBP > 185 or DBP > 110 unable to be treated with a continuous infusion, e.g., nicardipine);
14. Baseline CT/MR showing evidence of arterial vasculitis or dissection;
15. Baseline CT/MR evidence of multiple vascular territory acute stroke;
16. Excessive tortuosity of cervical vessels;
17. Intracranial stent in area that may impact Recanalization;
18. Presence of Pulmonary embolism, ilio-femoral or deep vein thrombosis
19. Presence of clinical signs of sepsis
20. Ongoing or spontaneous atrial fibrillation indicating severe peripheral vascular disease, aortic disease, or proximal cerebrovascular disease that in the opinion of the investigator precludes access or safe endovascular treatment
21. Presence of any other serious comorbidity that would be likely to impact life expectancy to less than 6 months or limit Patient cooperation or study compliance
22. Concurrent participation in an investigational clinical study (excluding registries) that has not completed the follow-up period or planned participation in another study within the next 3 months;
23. Patient has any other condition(s) or circumstance(s) that, in the judgement of the investigator, might interfere with or impact the collection of high quality data, or with the completion of follow up requirements within the study windows.
24. Patient has active or symptomatic COVID-19
25. Patients without a legally authorized representative to sign the consent form will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Test Arm patients achieving target temperature | 1 hour after thrombectomy
  Percentage of Test Arm patients achieving target temperature < 34 ºC within 1 hour of arterial puncture for thrombectomy
Mean door-to-Recanalization time | perioperative
  door-to-Recanalization time
Rate of hemorrhagic conversion in each arm within 36 hours of Recanalization | 36 hours
  Rate of hemorrhagic conversion

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Gupta, MD, MBA, Principal Investigator — Wellstar Medical Group
Locations (8):
- United States (8):
  - WellStar Kennestone Regional Medical Center, Marietta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Henry Ford, Detroit, Michigan
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Mercy Health, Toledo, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No